CLINICAL TRIAL: NCT02252484
Title: Energy Balance for Prostate Cancer Survivorship
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jill Hamilton-Reeves, PhD RD LD (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jill Hamilton-Reeves, PhD RD LD, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001274
Record Dates: First submitted 2014-09-18; First posted 2014-09-30 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostatectomy; weight loss; prevent weight gain
MeSH Terms: conditions — Prostatic Neoplasms; Weight Loss | interventions — Weight Reduction Programs; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight loss intervention Group (Experimental): Participants will receive tailor weight loss program. Participants will complete 8-weeks of the weight loss intervention prior to having their prostatectomy (weight loss phase). Program includes individual weight coaching, tailored diet and exercise plan, weight coaching and tracking of daily activities. Sessions will be held weekly during the weight loss phase. The groups will be facilitated by a registered dietitian with genitourinary (GU) oncology experience.
  Interventions: Other: Weight Loss Program
- Comparison Group (Active Comparator): All patients who are unwilling or not ready to engage in a weight loss program will be offered entry into the comparison group arm.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Weight Loss Program — Program has four main components: diet, physical activity, coaching and diet and exercise monitoring. The program is tailored to each individual in the study.
  Arms: Weight loss intervention Group
Other: Standard of Care — Standard of Care for this patient population.
  Arms: Comparison Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a weight management program for men undergoing a prostatectomy by seeing if the program is easy to follow, impacts weight gain, and reduces risk of cancer recurrence in the participants.

DETAILED DESCRIPTION:
The weight management program is designed to help participants lose weight before their prostatectomy and to help them maintain that weight loss after surgery. There are four main components to the weight management program. The four components of the program are:

1. Diet
2. Physical activity
3. Coaching
4. Diet and exercise monitoring tool

The program will be tailored to each individual participant. All participants will be ask to monitor their program using a tool provided by the study team. Participants will be actively participating in the study activities for about 5 months. After that, the study team will review medical records for up to 10 years after enrollment to monitor weight changes and cancer status.

ELIGIBILITY:
Inclusion Criteria:

* Men newly diagnosed with prostate cancer who are scheduled for prostatectomy (Stage T1 or T2)
* Body Mass Index (BMI) 25-45 kg/m2
* Have internet access
* Have an iPad/iPhone/iDevice

Exclusion Criteria:

* History of 5 alpha reductase inhibitors prior 3 months
* History of radiation therapy
* Taking active cancer treatment
* Undergoing salvage therapy
* Castration-resistant prostate cancer
* Evidence of metastasis
* Evidence of biochemical recurrence
* High risk medical condition (e.g. gout or kidney disease)

Ages: 50 Years to 72 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in body weight during the post-surgical period | Change from Surgery to Week 20

SECONDARY OUTCOMES:
Changes in body weight during the pre-surgical weight-loss intervention | Change from Baseline to Week 8
Changes in diet quality during the pre-surgical weight-loss intervention | Change from Baseline to Week 8
  Changes will be measured by analyzing results from alternative healthy eating index scores.
Prostate cancer status | Week 20
  Evidence of recurrence of cancer
Change in cardiovascular biomarkers | Change from Baseline to Week 20
  Changes will be measured by analyzing changes in participants lipid panel, c-reactive protein, fasting insulin and fasting glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Hamilton-Reeves, PhD, RD, LD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Derived] Hamilton-Reeves JM, Johnson CN, Hand LK, Bechtel MD, Robertson HL, Michel C, Metcalf M, Chalise P, Mahan NJ, Mirza M, Lee EK, Sullivan DK, Klemp JR, Befort CA, Parker WP, Gibbs HD, Demark-Wahnefried W, Thrasher JB. Feasibility of a Weight Management Program Tailored for Overweight Men with Localized Prostate Cancer - A Pilot Study. Nutr Cancer. 2021;73(11-12):2671-2686. doi: 10.1080/01635581.2020.1856890. Epub 2020 Dec 9. PMID 33295204